CLINICAL TRIAL: NCT00718120
Title: Immunogenicity and Safety Study of a Single Injection of GSK Biologicals' Trivalent Split Virion Influenza Vaccine Fluviral® (2008 - 2009 Season) in Adults Aged 18 to 60 Years and Over 60 Years.
Brief Title: Immunogenicity and Safety Study of GSK Biologicals' Fluviral® (2008 - 2009 Season) in Adults Over 18 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110584
Record Dates: First submitted 2008-07-17; First posted 2008-07-18 (Estimated); Results first posted 2009-08-25 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Influenza Vaccines
Keywords: Fluviral; Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

ARMS (2):
- Fluviral Adult Group (Experimental): Subjects aged between 18 and 60 years received a single dose of Fluviral® vaccine.
  Interventions: Biological: Fluviral®
- Fluviral Elderly Group (Experimental): Subjects aged more than 60 years received a single dose of Fluviral® vaccine.
  Interventions: Biological: Fluviral®

INTERVENTIONS:
Biological: Fluviral® — One intramuscular injection into the deltoid region of the non-dominant arm

SUMMARY:
This study will evaluate the immunogenicity and safety of GSK Biologicals' Trivalent split virion influenza vaccine Fluviral for the 2008-2009 season in adults over the age of 18.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* Male and female adults, 18 to 60 years of age and over 60 years of age.
* Written informed consent obtained from the subject.
* Satisfactory baseline medical assessment by history and physical examination.
* Comprehension of the study requirements, ability to comprehend and comply with procedures for collection of safety data, expressed availability for the required study period, and ability and willingness to attend scheduled visits.

Exclusion Criteria:

* Acute disease at the time of enrollment.
* Significant acute or chronic, uncontrolled medical or psychiatric illness.
* Any confirmed or suspected immunosuppressive condition including:

  * History of human immunodeficiency virus (HIV) infection,
  * Cancer or treatment for cancer, within 3 years of study enrollment. Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible.
* History of renal impairment.
* History of hepatic dysfunction due to hepatitis B, C or toxins including alcohol.
* Complicated insulin-dependent diabetes mellitus.
* Unstable cardiopulmonary disease requiring chronic medical therapy or associated with functional impairment.
* Presence of blood dyscrasias, including hemaglobinopathies and myelo- or lymphoproliferative disorder.
* Receipt of systemic glucocorticoids within 1 month of study enrollment, or any cytotoxic or immunosuppressive drugs within six months of study enrollment. Inhaled and topical steroids are allowed.
* A history of any demyelinating disease including Multiple Sclerosis and Guillain-Barré syndrome.
* Presence of an active neurological disorder.
* History of chronic alcohol consumption and/or drug abuse.
* Any significant disorder of coagulation that increases the risk of intramuscular injections or treatment with coumadin derivatives or heparin. Persons receiving prophylactic antiplatelet medications, e.g. low-dose aspirin, and without a clinically-apparent bleeding tendency are eligible.
* Receipt of an influenza vaccine within 6 months prior to study enrollment.
* Administration of any vaccines within 30 days prior to study enrollment or during the study period.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the vaccination or planned use during the study period.
* Administration of immunoglobulins and/or any blood products within the three months preceding the administration of the study vaccine or planned during the study.
* Any known or suspected allergy to any constituent of the vaccine.
* A history of severe adverse reaction to a previous influenza vaccination.
* If the subject is female, she must be of non-childbearing potential, or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for the duration of the study.
* Lactating/nursing female.
* Any condition which, in the opinion of the investigator, prevents the subject from participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2008-07-18 (Actual); Primary Completion 2008-08-09 (Actual); Study Completion 2008-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 110584 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110584 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110584 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110584 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110584 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110584 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110584 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group
Started | 55 | 55
Completed | 55 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (12.16) | 66.4 (4.61) | 53.2 (16.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 35 | 71
  Male | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Hemagglutination Inhibition (HI) Antibody Titers
Description: Titers, given as geometric mean titers (GMTs), are presented for all three vaccine influenza virus strains.
Time Frame: At Day 0 and 21
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group
Number analyzed (Participants) | 55 | 55
titer
  A/Brisbane (H1N1) [Day 0] | 19.5 [13.8 to 27.5] | 13.9 [10.7 to 18.2]
  A/Brisbane (H1N1) [Day 21] | 116.0 [88.4 to 152.2] | 47.1 [33.0 to 67.2]
  A/Uruguay (H3N2) [Day 0] | 19.1 [12.9 to 28.3] | 23.2 [16.0 to 33.8]
  A/Uruguay (H3N2) [Day 21] | 244.0 [173.5 to 343.2] | 170.3 [118.2 to 245.3]
  B/Florida [Day 0] | 59.8 [42.1 to 85.0] | 51.4 [36.3 to 72.8]
  B/Florida [Day 21] | 485.0 [378.9 to 620.8] | 256.6 [195.7 to 336.4]

2. Primary Outcome: Number of Seroconverted Subjects
Description: Seroconversion, defined as a pre-vaccination serum HI titer < 1:10 and a post-vaccination serum HI titer ≥ 1:40, or a pre-vaccination serum HI titer ≥ 1:10 and at least a 4-fold increase in post-vaccination serum HI titer, is presented for all three vaccine influenza virus strains.
Time Frame: At Day 21
Measure: Number; unit: subjects
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group
Number analyzed (Participants) | 55 | 55
subjects
  A/Brisbane (H1N1) | 28 | 18
  A/Uruguay (H3N2) | 40 | 35
  B/Florida | 38 | 25

3. Primary Outcome: Number of Seroprotected Subjects
Description: Seroprotection, defined as a serum HI antibody titer ≥ 1:40, is presented for all three vaccine influenza virus strains.
Time Frame: At Day 0 and 21
Measure: Number; unit: subjects
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group
Number analyzed (Participants) | 55 | 55
subjects
  A/Brisbane (H1N1) [Day 0] | 21 | 15
  A/Brisbane (H1N1) [Day 21] | 52 | 36
  A/Uruguay (H3N2) [Day 0] | 21 | 20
  A/Uruguay (H3N2) [Day 21] | 53 | 50
  B/Florida [Day 0] | 36 | 37
  B/Florida [Day 21] | 55 | 55

4. Primary Outcome: Fold Increase From Baseline in Serum HI Antibody Titer
Description: The fold increase in serum HI antibody titer post-vaccination (Day 21) compared to pre-vaccination (Day 0) was calculated by dividing the geometric mean antibody titers of Day 21 by those of Day 0. Data are presented for all three vaccine influenza virus strains.
Time Frame: At Day 21
Measure: Number; unit: fold increase
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group
Number analyzed (Participants) | 55 | 55
fold increase
  A/Brisbane (H1N1) | 6.0 | 3.4
  A/Uruguay (H3N2) | 12.8 | 7.3
  B/Florida | 8.1 | 5.0

5. Secondary Outcome: Number of Subjects Reporting Solicited Symptoms
Description: Solicited local symptoms assessed include pain, redness, and swelling. Solicited general symptoms assessed include bronchospasm, chills, cough, fatigue, headache, joint pain at other location, muscle aches, red eyes, sore throat, swelling of the face, and fever.
Time Frame: During the 4-day (Day 0-3) post-vaccination period
Measure: Number; unit: subjects
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group
Number analyzed (Participants) | 55 | 55
subjects
  Pain | 36 | 13
  Redness | 0 | 0
  Swelling | 2 | 0
  Bronchospasm | 1 | 2
  Chills | 2 | 0
  Cough | 1 | 4
  Fatigue | 10 | 8
  Headache | 14 | 6
  Joint pain at other location | 5 | 6
  Muscle aches | 19 | 11
  Red eyes | 3 | 4
  Sore throat | 7 | 3
  Swelling of the face | 0 | 0
  Fever | 1 | 0

6. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AE)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: During the 21-day (Day 0-20) post-vaccination period
Measure: Number; unit: subjects
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group
Number analyzed (Participants) | 55 | 55
subjects | 9 | 8

7. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAE)
Description: An SAE is any untoward medical occurrence that: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: During the 21-day (Day 0-20) post-vaccination period
Measure: Number; unit: subjects
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group
Number analyzed (Participants) | 55 | 55
subjects | 0 | 1

ADVERSE EVENTS:
Time Frame: Solicited adverse events were collected during the 4-day (Day 0-3) post-vaccination period, unsolicited and serious adverse events collected during the 21-day (Day 0-20) post-vaccination period.
Description: For this study, the Total Number (#) of Participants Affected by Other (non-serious) Adverse Events (AEs) was analyzed separately for expected AEs and for unexpected AEs. A consolidated analysis of all expected and unexpected AEs was not technically possible to be performed and the relevant data are no longer available. Therefore, the Total #Participants Affected in Other Adverse Events Table is currently populated by the highest value of #Participants affected within other AE's table.
Arm/Group | Fluviral Adult Group | Fluviral Elderly Group
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 1/55
Other Adverse Events (participants affected / at risk) | 36/55 | 13/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluviral Adult Group (N=55) | Fluviral Elderly Group (N=55)
Anaphylactic reaction (Immune system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluviral Adult Group (N=55) | Fluviral Elderly Group (N=55)
Cough (General disorders) | 1 | 4
Fatigue (General disorders) | 10 | 8
Headache (General disorders) | 14 | 6
Joint pain at other location (General disorders) | 5 | 6
Muscle aches (General disorders) | 19 | 11
Red eyes (General disorders) | 3 | 4
Sore throat (General disorders) | 7 | 3
Pain at the injection site (General disorders) | 36 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.